CLINICAL TRIAL: NCT03041870
Title: Relationship Between Serotonin and Brain Response to Social Dominance Perception and Emotion: a Combined [11C]DASB-PET/fMRI Study in Humans
Brief Title: Relationship Between Serotonin and Brain Response to Social Dominance and Emotion Perception.
Acronym: SERODOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL16_0014; 2016-A01588-43 (Other: ID-RCB)
Record Dates: First submitted 2017-01-31; First posted 2017-02-03 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Healthy Volunteers
Keywords: PET-fMRI; dominance; 5HT transporter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dominance (Experimental): Healthy subjects
  Interventions: Device: PET-fMRI scan

INTERVENTIONS:
Device: PET-fMRI scan — fMRI scan include MR sequences: BOLD and fMRI. The PET acquisition will be carried out in dynamic for 90 consecutive minutes following intravenous administration of 4 MBq / kg dose of [11C]DASB bolus.

SUMMARY:
Previous studies have already revealed the involvement of the serotoninergic system in the social behavior process. For example, more serotonin (5HT) was found in dominant male adult monkeys. Little is known about the serotoninergic implication in human's social behavior. The project aims to clarify the role of the serotoninergic system in social behavior in relation to the process of social hierarchical information. In order to determine how serotoninergic system is involved, the investigator will use a new technic TEP-fMRI. This technic allows us to measure the brain activity and the serotoninergic transporter occupancy (using the [C11]-DASB) at the same time. The current study aims to investigate whether serotonin transporter (5-HTT) activity correlates with the neural response (BOLD) during the detection of social dominance in facial expressions or other measures of social information processing. Blood sample, SLC6A4 (allele coding for the 5HT transporter) genotyping and neuropsychological questionnaires will give at the investigator more information and allow to investigate whether performance on social information processing is modulated by personality trait and genotype.

ELIGIBILITY:
Inclusion Criteria:

* French speaking
* Normal vision
* Age from 18 to 45
* Without psychiatric antecedent
* Without any neurologic antecedent
* Not taking psychotropic or anxiolytic drugs
* Having health insurance coverage

Exclusion Criteria:

* The subject does not wish to be notified of any anomalies detected during MRI
* Subjects suffering from claustrophobia
* Subjects carrying magnetic metal objects that cannot be removed as cochlear implant, surgical clips, piercings, pacemakers, mechanical valves
* Subjects participating in a clinical trial or being in a period of exclusion from a previous clinical trial
* Person under guardianship or curatorship or deprived of liberty or in emergencies
* Taking unauthorized treatment in the month before the completion of the review
* Person whose physical or mental condition does not allow him to pass the test study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
level of Blood-Oxygen-Level Dependent (BOLD) signal | at day 0
  The BOLD signal will be measured using a MRI scanner, and simultaneously we will record the level of serotonin transporter with [11C]DASB marker of the serotonin transmission, using a PET signal. We will use the Scatchard method in order to determine the level of [11C]DASB bonded to the transporter. Our reference region will be the cerebellum.
level of serotonin transporter | at day 0
  The BOLD signal will be measured using a MRI scanner, and simultaneously we will record the level of serotonin transporter with [11C]DASB marker of the serotonin transmission, using a PET signal. We will use the Scatchard method in order to determine the level of [11C]DASB bonded to the transporter. Our reference region will be the cerebellum.

SECONDARY OUTCOMES:
Behavioral assessment | at day 0
  During the entire scanner, subjects will be ask to perform a behavioral task. Their responses will be analyzed.
Testosterone Blood level | after the scan session at day 0
  The testosterone will be measured on a blood sample.
Cortisol Blood level | after the scan session at day 0
  The cortisol will be measured on a blood sample (prelevated at same time than testosterone).
SLC6A4 genotyping | at day 0
  The genotyping of this gene (SLC6A4) will be realized on a sample of saliva.

CONTACTS AND LOCATIONS:
Overall Officials: Christian SCHEIBER, Principal Investigator — Hospices Civils de Lyon - CNRS UMR 5229
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No